CLINICAL TRIAL: NCT06159556
Title: Effect of Daily Consumption of Peanuts on Immune Function and Cardiometabolic Markers and Risk Factors in Free-living Individuals: A Randomized Controlled Trial
Brief Title: Effects of Peanuts on Immunity and Cardiometabolic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5230190
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Immune Response; Cardiometabolic Risk Factors
Keywords: Peanuts; Immunity; heart disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: The proposed study is a 12 week parallel- group , free living, observer-blind randomized controlled study with 80 adult men and women
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor will not be aware which participant is in what arm. The participant and the care provider will know about the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut group (Active Comparator): Participants will be consuming 2 ounces of peanuts /peanut butter everyday for 12 weeks
  Interventions: Other: Peanut intake
- control group (No Intervention): Participants will continue with habitual diet and abstain from eating peanuts

INTERVENTIONS:
Other: Peanut intake — Participants will consume 2 ounces of peanuts/peanut butter for 12 weeks
  Arms: Peanut group

SUMMARY:
The aim of the proposed study is two-fold: to determine whether the intake of peanuts (a) enhances immune function and (b) produces a desirable impact on selected cardiometabolic biomarkers and risk factors.

DETAILED DESCRIPTION:
The aim of the proposed study is two-fold: to determine whether the intake of peanuts (a) enhances immune function and (b) produces a desirable impact on selected cardiometabolic biomarkers and risk factors . To accomplish this objective, a human dietary intervention trial (RCT) with peanuts is proposed. The proposed study is a 12-week parallel-group, free-living, observer-blind, randomized controlled dietary intervention trial. This study will examine the effects of peanuts on markers of immune function, cardiometabolic markers and risk factors and upper respiratory tract infections, in 80 adult male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* adults between the ages of 18-70 years

Exclusion Criteria:

* known intolerance or allergy to peanuts
* bad dentures unable to chew peanuts
* regular intake of peanuts and/or other nuts (>3 ounces/week)
* use of immune-boosting supplements
* exposure to antibiotics and corticoids immediately prior to the study
* use of other medications or supplements that can interfere with the immune functions
* Individuals that received any vaccination (i.e flu or Covid 19) 6 months prior to the start of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Changes in lymphocyte populations | baseline to 12 weeks
  Immunophenotyping will be performed by flow cytometry to measure the number of T helper, T cytotoxic, Naive and memory cells and B cells
Changes in Lymphocyte activity | baseline to 12 weeks
  The production of lymphocytes will be measured in the supernatant using enzyme linked immunosorbent assay (ELISA)
Changes in cytokine production | baseline to 12 weeks
  The cytokines produced due to lymphocyte activity will be measured in the supernatant using enzyme linked immunosorbent assay (ELISA)
Changes in serum inflammatory cytokine concentration | baseline to 12 weeks
  changes in the concentrations of the inflammatory cytokines will be performed on serum using enzyme linked immunoassay (ELISA) will include hs-CRP, interleukin (IL)-1B, IL-6, TNF a, IL-10 and IFN-γ, MCP1, Eotaxin, E-selectin, RANTES and Pentraxin-3
Changes in the serum lipid concentration | baseline to 12 weeks
  This is a composite measurement which will measure the changes in the levels of serum low density cholesterol, high density cholesterol, non- high density cholesterol and triglycerides
Changes in insulin resistance | baseline to 12 weeks
  Change in insulin resistance will be measured using the Hemostatic Model Assessment calculator version 2 (HOMA2-IR)
Changes in Hemoglobin A1c | baseline to 12 weeks
  Change in Hemoglobin A1c will be measured by cation-exchange high-performance liquid chromatography method
Changes in body weight | baseline to 12 weeks
  A change in body weight for both the peanut and control group will be measured using an In Body machine at the baseline and end of intervention
changes in systolic and diastolic blood pressure | baseline to 12 weeks
  Seated systolic and diastolic blood pressure will be measured at baseline and end of intervention utilizing Omron -Model HEM-7471 C device. Three measurements will be taken after a five-minute rest period, 1 minute apart, and the last two recordings will be averaged for analysis.
changes in percentage body fat | baseline to 12 weeks
  A change in the percentage of body fat for both the peanut and control group will be measured using an In Body machine at the baseline and end of intervention

SECONDARY OUTCOMES:
changes in upper respiratory infection questionnaire score | baseline to 12 weeks
  Upper respiratory tract infections will be tracked using the Jackson and Dowling questionnaire. The questionnaire will be completed daily by participants, either manually or electronically , throughout the 12-week study period. The scale for the questionnaire is from 0-42. The higher score means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No